CLINICAL TRIAL: NCT01628003
Title: Study of Reserves After Traumatic Brain Injury:Influence of Brain, Cognitive, and Emotional Reserves on Long-Term Consequences of Traumatic Brain Injury
Brief Title: Study of Reserves After Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-09-7297-AS-CTIL
Record Dates: First submitted 2012-06-19; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; long-term outcome; Brain Reserves; Cognitive Reserves; Emotional Reserves; Patients 1 year or more after Moderate or Severe Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy persons (Active Comparator)
  Interventions: Device: Brain MRI; Device: MRI
- patients after moderate-severe TBI (Experimental)
  Interventions: Device: Brain MRI; Device: MRI

INTERVENTIONS:
Device: Brain MRI — Brain MRI
Device: MRI — Physical examination Neuropsychological testing Questionnaires

SUMMARY:
It is hypothesized that the long-term results of rehabilitation and subsequent aging after Brain Trauma depend on brain's premorbid anatomical (structural) and functional (cognitive, emotional) reserves.

The purpose of this study are:

1. to determine whether such reserves exist.
2. to study their convergent and discriminant validity.
3. to study their characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-Severe Traumatic Brain Injury according to at least 1 the following:

  * Duration of loss of consciousness (LOC) - more then 1/2 hour
  * Glasgow Coma Scale (GCS) - less then 13
  * Post Traumatic Amnesia (PTA) - more then 24 hours.
* At least 1 year after the injury.

Exclusion Criteria:

* Mild Traumatic Brain Injury
* the present state of Post Traumatic Amnesia
* dementia
* the age less than 18 years on the moment of injury
* less than 1 year since the injury
* incapacity of the patient to cooperate in the study (incapacity of any source including physical, mental, and language problems)
* premorbid diagnosis of Mental Retardation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological battery | neuropsychological baterry for every participant will be performed during 3-4 meetings. An expected average for complete neuropsychological assessment is about 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Tel Hashomer Medical Center, Ramat Gan, Israel